CLINICAL TRIAL: NCT05721469
Title: The Effect of Art Therapy Applied to Mothers on Eating Behavior in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif AKYİĞİT ALBAYRAK, Lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 78794538
Record Dates: First submitted 2022-12-29; First posted 2023-02-10 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Art Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled pretest posttest applied art therapy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kontrol group (No Intervention): Pretest and posttest application
- experimental group (Experimental): Art therapy application to the experimental group
  Interventions: Behavioral: Art therapy
- Posttest phase (No Intervention): Applying posttest to the experimental and control groups

INTERVENTIONS:
Behavioral: Art therapy — Determining the mothers of children with eating disorders with the data obtained from the questionnaires and scales and separating them into randomized experimental and control groups, 8-12 sessions of 90 minutes of music, painting, ceramics, etc. were given to the mothers participating in the experimental group. Art Therapy Studies
  Arms: experimental group

SUMMARY:
Art therapy; Art therapy is an integrative mental health service that enriches the lives of individuals, families, and communities through active art practices, the creative process, applied psychological theory, and human experience in a psychotherapeutic relationship. It is a therapeutic method used in the form of sessions to improve self-esteem and self-esteem." Art therapy used to develop emotional resilience, increase insight, develop social skills, reduce and resolve conflicts and distress seeks to both find an outlet for complex and intense emotions and It allows them to be verbally expressed at an intellectual level, and aims to develop and grow self-awareness within themselves.

DETAILED DESCRIPTION:
Art Therapy, a term that has its origins in art and psychotherapy, was first used by Adrian Hill in the 1940s in the treatment of tuberculosis patients, and then it began to be used in cancer and post-traumatic stress disorder. In this process, these people needed less medication and it was determined that the patients experienced less loneliness. In parallel with today's social developments, the changing needs of individuals and communities also affect the view of health, and today, a health-centered care approach that protects, maintains and improves the health of the individual, family and society comes to the fore . In this context, art therapy is applied by trained art therapists and/or practitioners in many of the health care fields such as dance/movement therapy, drama therapy, music therapy, poetry therapy and psychodrama therapy, and it has been proven by various studies that positive results are obtained in treatment processes.

Art therapy, together with music and dance, is seen as a component of complementary medicine and is seen as a treatment method in the management of many mental and non-psychological pathological or nonpathological conditions. In a study conducted by Raybin and Krajicek on the application of art therapy in children with cancer, it was stated that the quality of life in children increased, children felt better, psychosocial symptoms decreased, and cancer-related pain was felt less after art therapy applications. In another study; 78 children between the ages of 3 and 11 who were to undergo general anesthesia before the operation were allocated to the experimental and control groups, general anesthesia was applied to the control group after the standard application, and integrated art therapy and clown visits were made to the experimental group for a while when they came to the hospital and before the operation. When children in the experimental group were compared with those in the control group, a significant decrease was found in the Modified Yale Preoperative Anxiety Scale scores in case of separation from their parents. In addition, most of the parents and nurses stated that it was effective in reducing the anxiety of the children in the experimental group.

In a pretest-posttest quasi-experimental study examining the effect of art psychotherapy using marbling; Volunteer participants exposed to domestic violence were subjected to marbling practice for 14 weeks, interviews were conducted with psychotherapy methods and therapeutic cooperation, and after these interviews, it was determined that the participants' Beck Depression Scale and Anxiety and Hopelessness Scales Questionnaire scores were lower than their pretest scores . Regarding Eating Behavior in Children; Feeding and eating difficulties, which can be seen very often, are accepted as part of abnormal development. It is known that many parents talk about many conditions such as undereating or overeating, fast or slow eating, etc. of their children. These conditions may be a precursor to a disease of clinical importance. These problems, which initially appear as eating problems, can then progress to a more difficult process in the form of refusal to eat, overeating or weight loss difficulties. In a study conducted; Thirty adolescents with Anorexia Nervosa and Obsessive Compulsive features received 15 sessions of family-based therapy and cognitive enhancement therapy (15 adolescents) and family-based therapy and art therapy . Adolescents and family-based treatment and cognitive improvement therapy group, moderate changes were found in cognitive disabilities, whereas it was reported that there was a high and significant change in cognitive level in patients who received family-based treatment and art therapy.

In a study on music therapy, Wang and Agius stated that Music Therapy is effective on Depression, Anxiety, Schizophrenia, Sleep Disorders and Dementia, and patient participation is required to increase this effect. Wigham et al. In a systematic review they have done; They stated that art therapy applied to children with long-term physical problems had some positive developments in children's mental health and well-being indicators, including quality of life, coping behaviors, anxiety, self-concept and mood. emphasized In a qualitative study; Open-ended, structured interviews were conducted with parents of children with eating disorders, and they stated that they felt guilty about the disease, and that they had problems in coping with the health problems that resulted from eating disorders in their children. As a result of the interviews conducted in the study, they mentioned that progress has been made in coping methods such as hope, optimistic thinking, never giving up, and determination, and as a result of the findings, parents of children with eating disorders should be educated within the scope of health care. In the study, it was stated that the parents of children with eating disorders lacked interest in their children and emphasized the importance of family involvement in the treatment of eating disorders.

In another study; As a result of 90-minute psychoeducational meetings with the parents of children with eating disorders, it was observed that the emotional functioning levels of the parents increased, their feelings of guilt and shame decreased, and there were significant changes in their behavior towards their children with eating disorders .

When the studies conducted in recent years are examined, it is seen that the application area of art therapy is not one-sided, Autism Spectrum Disorder, Down Syndrome, Learning Disorder, etc. It has also been proven that it has positive effects on individuals with many physical and mental illnesses, the people responsible for their care, and nurses .

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years or older
* Having a child who continues pre-school education

Exclusion Criteria:

* The mothers included in the study quit the study,
* Having problems in repeating the methods to be applied in art therapy,
* Does not accept home visits,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is aimed at women, as the mother's effect on eating behavior and women's empowerment are examined.
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Identifying the eating behavior problem | 4 month
  The Feeding Process Mother Attitudes Scale will be used to determine eating problems in the pretest phase.
Identifying coping strategies | 4 month
  The Coping Strategies Short Form will be used in the pre-test phase.
Practicing art therapy | 4 month
  Eating behavior changes in children by applying art therapy,

CONTACTS AND LOCATIONS:
Overall Officials: Elif Akyiğit Albayrak, Principal Investigator — Hasan Kalyoncu Universty Gaziantep,Turkey
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No